CLINICAL TRIAL: NCT05435833
Title: Ultrasound-Guided Submandibular Parapharyngeal Glossopharyngeal Nerve Block for Post -Tonsillectomy Pain Relief in Adults. A Prospective Randomized Study
Brief Title: Glossopharyngeal Nerve Block for Post -Tonsillectomy Pain Relief
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Gehan Morsy Eid (Unknown); Aliaa Muhammad Belal (Unknown); Mohamed Shebl Abdelghany (Unknown)
Responsible Party: Principal Investigator, Mona Blough El Mourad, Assistant professor of Anesthesia, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GPN block in tonsillectomy
Record Dates: First submitted 2022-06-18; First posted 2022-06-28 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (glossopharyngeal nerve block group) (Experimental): bilateral ultrasound guided GPN block will be performed after induction of anesthesia and pre incisional by an experienced anesthesiologist
  Interventions: Procedure: bilateral ultrasound guided GPN block
- Group II(Control group) (No Intervention): general anesthesia alone (no block)

INTERVENTIONS:
Procedure: bilateral ultrasound guided GPN block — a linear high frequency ultrasound probe will be initially positioned over the hyoid bone in the transverse plane, then the probe will be rotated to keep in line with the mandibular angle and the pharyngeal wall is identified by US. Using an in plane approach, a 22 G ,5 cm needle will be advanced till it reaches just superficial to the pharyngeal wall and 2.2 ml of 0.25% bupivacaine will be injected.
  Arms: Group I (glossopharyngeal nerve block group)

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of Ultra-sound guided submandibular parapharyngeal glossopharyngeal nerve block as regards time for first need of analgesic as a primary outcome as well as pain score, total postoperative analgesic requirement, and incidence of complications as secondary outcomes

DETAILED DESCRIPTION:
Tonsillectomy is one of the most frequent surgical procedures performed all over the world that has been identified as being severely painful especially in the adult population. Management of post tonsillectomy pain is of paramount importance in order to improve swallowing and enhance oral intake as well as to decrease the risk of dehydration, infection and secondary hemorrhage with a subsequent hastening of recovery.

A variety of analgesic regimens have been implemented to alleviate post-tonsillectomy pain, however; no consensus on the ideal analgesic regimen has been yet identified.

The Ultrasound (US)-guided glossopharyngeal nerve (GPN) block has been acknowledged as a feasible option for providing perioperative analgesia in tonsillectomy patients. It blocks sensory impulses from the posterior third of the tongue, palatine tonsil, and mucous membranes of the mouth and pharynx. Conventional techniques for blocking the GPN carry the risk of vascular puncture, inadvertent block of closely adjacent other cranial nerves, with increased probability of local anesthetic toxicity and even upper airway obstruction. Recently, a novel, safe, and reproducible US-guided GPN block technique has been introduced by Azman et al, which would block the GPN distally, in the tissue plane just next to the pharyngeal wall and relatively far from high risk nearby structures.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified by the American society of Anesthesiologists ASA I and II patients
* Scheduled for tonsillectomy procedure

Exclusion Criteria:

* Patients' refusal
* History of diabetes mellitus,
* Cardiac, liver or renal impairment
* Obstructive sleep apnea syndrome
* Swallowing difficulty
* Intake of chronic pain medications or substance abuse
* Bleeding disorders
* Hypersensitivity to the used medication

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Onset of 1st analgesic request | up to 24 hours postoperative
  the time to first analgesic request will be recorded

SECONDARY OUTCOMES:
Pain score | at 30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours postoperative
  The numerical rating scale for pain ranging from 0-10 where the minimum value of 0 represents no pain and the maximum value of 10 represent the worst pain imaginable
Postoperative rescue analgesic consumption | up to 24hours postoperative
  Total 24 hours postoperative rescue analgesic consumption

CONTACTS AND LOCATIONS:
Overall Officials: Mona B El Mourad, MD, Principal Investigator — Tanta University
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Kim MS, Choi HG, Park EK, Kim SY, Kim JH, Park B. Natural course of tonsillectomy pain: A prospective patient cohort study. Auris Nasus Larynx. 2018 Jun;45(3):508-513. doi: 10.1016/j.anl.2017.07.018. Epub 2017 Sep 8. PMID 28890114
- [Background] Ahmed SA, Omara AF. The Effect of Glossopharyngeal Nerve Block on Post-Tonsillectomy Pain of Children; Randomized Controlled Trial. Anesth Pain Med. 2019 Apr 30;9(2):e90854. doi: 10.5812/aapm.90854. eCollection 2019 Apr. PMID 31341828
- [Background] Ozalevli M, Unlugenc H, Tuncer U, Gunes Y, Ozcengiz D. Comparison of morphine and tramadol by patient-controlled analgesia for postoperative analgesia after tonsillectomy in children. Paediatr Anaesth. 2005 Nov;15(11):979-84. doi: 10.1111/j.1460-9592.2005.01591.x. PMID 16238560
- [Background] Naesh O, Niles LA, Gilbert JG, Ammar MM, Phibbs PW, Phillips AM, Khrapov AV, Robert AJ, McClintock A. A randomized, placebo-controlled study of rofecoxib with paracetamol in early post-tonsillectomy pain in adults. Eur J Anaesthesiol. 2005 Oct;22(10):768-73. doi: 10.1017/s0265021505001274. PMID 16211736
- [Background] Hanasono MM, Lalakea ML, Mikulec AA, Shepard KG, Wellis V, Messner AH. Perioperative steroids in tonsillectomy using electrocautery and sharp dissection techniques. Arch Otolaryngol Head Neck Surg. 2004 Aug;130(8):917-21. doi: 10.1001/archotol.130.8.917. PMID 15313860
- [Background] Kaygusuz I, Susaman N. The effects of dexamethasone, bupivacaine and topical lidocaine spray on pain after tonsillectomy. Int J Pediatr Otorhinolaryngol. 2003 Jul;67(7):737-42. doi: 10.1016/s0165-5876(03)00091-0. PMID 12791448
- [Background] Ginstrom R, Silvola J, Saarnivaara L. Local bupivacaine-epinephrine infiltration combined with general anesthesia for adult tonsillectomy. Acta Otolaryngol. 2005 Sep;125(9):972-5. doi: 10.1080/00016480510043413. PMID 16193589
- [Background] Aldamluji N, Burgess A, Pogatzki-Zahn E, Raeder J, Beloeil H; PROSPECT Working Group collaborators*. PROSPECT guideline for tonsillectomy: systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Jul;76(7):947-961. doi: 10.1111/anae.15299. Epub 2020 Nov 17. PMID 33201518
- [Background] Tolska HK, Hamunen K, Takala A, Kontinen VK. Systematic review of analgesics and dexamethasone for post-tonsillectomy pain in adults. Br J Anaesth. 2019 Aug;123(2):e397-e411. doi: 10.1016/j.bja.2019.04.063. Epub 2019 Jun 17. PMID 31221427
- [Background] Sirohiya P, Kumar V, Yadav P, Bharti SJ. Ultrasound-Guided Glossopharyngeal Nerve Block at Pharyngeal Wall Level in a Patient with Carcinoma Tongue. Indian J Palliat Care. 2020 Jan-Mar;26(1):140-141. doi: 10.4103/IJPC.IJPC_132_19. Epub 2020 Jan 28. PMID 32132800
- [Background] Manoharan D, Bharati SJ, Yadav MK. A novel technique of ultrasound-guided glossopharyngeal nerve block to relieve cancer pain. Saudi J Anaesth. 2019 Jul-Sep;13(3):279-280. doi: 10.4103/sja.SJA_139_19. No abstract available. PMID 31333392
- [Background] Bean-Lijewski JD. Glossopharyngeal nerve block for pain relief after pediatric tonsillectomy: retrospective analysis and two cases of life-threatening upper airway obstruction from an interrupted trial. Anesth Analg. 1997 Jun;84(6):1232-8. doi: 10.1097/00000539-199706000-00011. PMID 9174298
- [Background] Azman J, Stopar Pintaric T, Cvetko E, Vlassakov K. Ultrasound-Guided Glossopharyngeal Nerve Block: A Cadaver and a Volunteer Sonoanatomy Study. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):252-258. doi: 10.1097/AAP.0000000000000561. PMID 28195898